CLINICAL TRIAL: NCT04493723
Title: Molecular Characterisation of Serial Tumour Samples and Their Correlation With Circulating Biomarkers and Other Biospecimens Taken During the Clinical Course of Patients Receiving Treatment for Malignant Melanoma.
Brief Title: Serial Tumour Biopsies and Blood Biomarkers in Melanoma
Status: Recruiting | Type: Observational
Sponsor: The Christie NHS Foundation Trust (Other)
Collaborators: University of Manchester (Other)
Responsible Party: Sponsor
Other Study IDs: CFTSp157; 18/NW/0515 (Other: Preston NW REC); 132792 (Other: IRAS)
Record Dates: First submitted 2020-07-21; First posted 2020-07-30 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Melanoma
Keywords: Tumour Biopsy; Blood Biomarker
MeSH Terms: conditions — Melanoma | interventions — Surgical Procedures, Operative; Biopsy; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Tumour biopsies, whole blood and blood products
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All participants: All eligible, consented participants, will be asked to give blood, tissue, and other biospecimens for research purposes
  Interventions: Procedure: Surgery; Procedure: Venepuncture

INTERVENTIONS:
Procedure: Surgery — To collect tumour tissue
  Other Names: Biopsy
Procedure: Venepuncture — To collect blood samples

SUMMARY:
Recent advances in understanding how cancer develops and spreads have led to effective new treatments and improved outcomes for patients with melanoma. However, we know that these new treatments do not work for all patients: some do not respond to them and some initially respond but then develop resistance. The overall aim of this study will be to collect tumour biopsies, biomarkers present in the blood, and other biological specimens which can be used to try to understand why resistance to anti-cancer treatment occurs, and to develop predictive biomarkers of this resistance in patients with locally advanced and metastatic malignant melanoma.

The study will be open to NHS patients aged 16 and over, who have been diagnosed with advanced melanoma, and who will be receiving treatment for their disease as part of their routine care. Patients will be asked to provide samples from tumour biopsies before, during and after treatment. We will also ask for blood samples to look at biomarkers in the blood and see how these correspond with tumour samples, which will further help us to understand treatment response. Biomarkers are substances in the body that can be measured and help indicate how a disease is developing. It is hoped that soon we will be able to monitor cancer by analysing a patient's blood samples, thus reducing the need for biopsies. As blood tests could be taken more frequently, signs that patients are becoming resistant to treatments could be picked up sooner.

As well as monitoring biomarkers, we would also like to understand what happens to the healthy cells surrounding the tumour during treatment. This will improve our understanding of how cells adapt and respond to treatments, and may eventually lead to the discovery of new biomarkers to help predict which patients will develop resistance to certain treatments.

DETAILED DESCRIPTION:
This will be a prospective study recruiting patients who have been diagnosed wth advanced melanoma.

Participants will be asked to give informed consent before any samples are collected.

Participants will be asked to donate tissue and other biospecimens (see list below) that are surplus to clinical requirements if a participant is undergoing any of the following as part of their routine care:

* lymph node dissection
* sentinel lymph node biopsy as part of their normal care
* resection of metastatic skin lesions or visceral disease
* medical treatment for Stage IV disease Biospecimens include urine, stool, saliva, hair follicles, ascitic, pleural, pericardial or cerebrospinal fluid Collection of archival tumour tissue from previous biopsy/surgery that is surplus to clinical requirements will also be requested, where available.

Participants will be asked to consent to having easily accessible lesions biopsied or resected, which are not required for clinical reasons, but are for research purposes only. Participants can still be part of the study even if they do not agree to these extra, optional biopsies. Tissue samples from the surgical specimens and the original primaries will be examined to look for molecular markers to correlate with circulating tumour molecular markers.

Consent will be requested to grow cell lines from the donated tumour tissue and implant tumour tissue into mice to characterise the genetic changes seen in both CTCs and biopsies, in terms of resistance to targeted agents, in the lab setting. Consent to this part of the study will be optional.

A maximum of 50mls blood sample will be requested from participants before any intervention. Further blood samples (maximum of 50mls each time) will also be requested as follows:

* after surgery, on subsequent routine follow up at 3 months, and then 3 monthly thereafter (i.e. approximately 4 times in a year after the initial pre and post surgical specimens)
* at the time of disease recurrence
* If on treatment, then usually approximately 3 weeks after starting treatment, and then every 2 cycles of treatment
* at disease progression The samples will be tested for various circulating tumour biomarkers.

We will be asking a small group of patients, approx 20, to consent to weekly blood samples, for up to 8 weeks, for specific biomarker analyses.

Clinical data will be collected for each patient, looking at demographics, baseline haematology and biochemistry blood results, radiological extent of disease, time to disease progression, clinical and histological features of the primary. Patients will be followed up for approximately 10 years to assess their outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 16 years or more.
2. Patients must have given written informed consent.
3. Evidence of locally advanced or metastatic melanoma, i.e. stage III or IV disease.
4. Accessible tumour that can be safely biopsied using radiological or surgical techniques (if consenting to part A).
5. Full blood count and coagulation tests within acceptable parameters (if consenting to part A).

Exclusion Criteria:

1. Inability to provide informed consent.
2. History of significant bleeding disorder (patients on anticoagulation are eligible if the anticoagulation can be safely managed to allow fresh tumour biopsies and blood sampling).
3. History of HIV, Hepatitis B/C or other transmissible human disease.
4. Any conditions where research biopsies or blood sampling may increase risk of complications for the patient and/or investigator, including high risk groups such as intravenous drug users.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with stage III or IV melanoma undergoing systemic therapy at The Christie hospital
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-11-14 (Actual); Primary Completion 2034-07 (Estimated); Study Completion 2034-07 (Estimated)

PRIMARY OUTCOMES:
The number of patients who consent to have additional samples taken for research purposes and the number of research samples collected. | Duration of study, 300 participants over 16 years
  This is primarily a sample collection study, where tissue will be used in future experiments to further understand mechanisms of disease resistance. This study will however assess patients acceptability to enrol in a study, where biological samples are taken purely for research, and not part of routine care.

CONTACTS AND LOCATIONS:
Overall Officials: Lorigan, Prof, Principal Investigator — University of Manchester
Locations (1):
- The Christie, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plans to share IPD